CLINICAL TRIAL: NCT06815107
Title: Risk Factors for Poor Tolerance of Ureteral Double-J Stent
Acronym: ToleJJ
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Centre Hospitalier d'Abbeville (Other); centre hospitalier de Compiegne (Unknown); University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2020_843_0029
Record Dates: First submitted 2025-02-04; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Tolerance; Ureteral Double-J Stent; Urinary Symptoms
Keywords: Ureteral Double-J Stent; tolerance; urinary symptom

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: questionnary — On day 1 of an ureteral double J stenting, each participant will receive the first USSQ questionnaire, in the French validated version. This questionnaire will be completed at home, one week after the intervention and returned at the following consultation or hospitalization.
Other: USSQ survey — if the stent is removed less than 6 months later, the second USSQ survey, in the French validated version will be given to the patient when removing the stent. This questionnaire will be completed at home one week after removal of the stent and return to the referent hospital. If the patient does not return the second questionnaire, our team may contact them by phone to complete it.

SUMMARY:
The placement of a Ureteral Double-J Stent as an emergency treatment or preparation for endoscopy after Colic nephritis is very frequent. It is often poorly supported, most often by young patients. A rich symptomatology is related to the probe responsible for a limitation of activities that can have a strong socio-economic impact. The objective of this study is the identification of the predictive factors of poor tolerance.

ELIGIBILITY:
Inclusion Criteria:

* patient over 18 years old
* patient who need Ureteral Double-J Stenting

Exclusion Criteria:

* patient under 18 years old,
* Iterative change,
* understanding disorder,
* inability to answer the questionnaire,
* refusal of the patient,
* long-term Ureteral Double-J Stenting (more than 6 month),
* active cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-04-15 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
tolerance score of Ureteral Double-J Stent | day 15
  A tolerance score of Ureteral Double-J Stent will be established using the USSQ questionnaire allowing the comparison of the symptomatology with and after ablation of the stent
tolerance score of Ureteral Double-J Stent | 3 months
  A tolerance score of Ureteral Double-J Stent will be established using the USSQ questionnaire allowing the comparison of the symptomatology with and after ablation of the stent

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens-Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No